CLINICAL TRIAL: NCT03160651
Title: Corticosteroids in Severe Alcoholic Hepatitis Patients With Early Spontaneous Improvement
Brief Title: Corticosteroids in Alcoholic Hepatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORTISAVE study
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis; spontaneous improvement; corticosteroids
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind randomized trial Investigator, patients, and care providers will be masking Only statisticians and pharmacist will not be masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methylprednisolone (Active Comparator): Patients will receive 28 days of methylprednisolone 32 mg/day
  Interventions: Drug: Methylprednisolone or placebo
- placebo (Placebo Comparator): Patients will receive 28 days of matching placebo
  Interventions: Drug: Methylprednisolone or placebo

INTERVENTIONS:
Drug: Methylprednisolone or placebo — Patients will receive 28 days of methylprednisolone 32 mg/day

SUMMARY:
Approximately 50% of patients admitted for severe AH will have spontaneous improvement of liver function before initiation of therapy (ie decrease in mDF between hospital admission and initiation of steroids). These patients have a better prognosis than patients without spontaneous improvement of liver function. It has never been demonstrated that corticosteroids improve survival in severe AH patients with spontaneous improvement of liver function. Our hypothesis is that severe AH patients with spontaneous improvement of liver function represent a group who could most benefit from steroids

ELIGIBILITY:
Inclusion Criteria:

1. Clinical syndrome of alcoholic hepatitis:

   recent jaudice or in recent aggravation (< 3 months) serum bilirubin > 5 mg/dL history of excess alcohol abuse (> 40g/day)
2. Alcoholic hepatitis proven by a liver biopsy (histological criteria of alcoholic hepatitis defined according to EASL clinical practice guidelines : steatosis, hepatocyte ballooning, and an inflammatory infiltrate with PMNs). The results of the liver biopsy are not mandatory for inclusion. However, the biopsy must be planned at the latest on day 1. When the results become available and do not confirm alcoholic hepatitis, the patient must discontinue the study.
3. Spontaneous liver function improvement, defined by a decrease in serum bilirubin level > 10% between admission and day 5-10 after admission
4. less than 2 weeks since admission to hospital
5. Maddrey discriminant function* greater than or equal to 32
6. Subjects must voluntarily sign and date an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) prior to the initiation of any screening or study-specific procedures.
7. Subjects must be able to understand and adhere to the study visit schedule and all other protocol requirements.

Patients with significant hepatic encephalopathy are not excluded from participation to the trial. In this case, the patient should be accompanied by a legal representative that will decide participation in the clinical study and sign ICF.

Exclusion Criteria:

1. Other causes of liver disease including viral hepatitis (positive HBs antigen, HCV RNA positive), auto-immune hepatitis, biliary obstruction
2. Other disease compromising 90-day survival
3. Positive HIV serology
4. Uncontrolled infection All patients will be screened for infection. This will involve chest radiography, urinalysis, PMNs count in ascites (if ascites present). All other sign or clinical suspicion of infection with or without antibiotherapy will be recorded as an infection.

   Positive culture and initiation of antibiotics with clinical or radiological signs of infection, as well as clinical suspicion, will be recorded as infection.

   Patients with evidence of sepsis will be treated for a minimum of 2 days with appropriate antibiotics. Once the local principal investigator considers that the sepsis is under control, the patient may be rescreened and randomised.
5. Uncontrolled gastrointestinal bleeding Bleeding must be judged as controlled for at least 5 days
6. Patient with serum creatinine > 2.5 mg/dL, under renal replacement therapy or under terlipressine (or other vasoactive drugs)
7. Pentoxyphilline therapy
8. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mortality at 90 days | 90 days
  To determine whether Methylprednisolone compared to placebo improve the 90 day mortality from patients with severe AH and spontaneous improvement of liver function

SECONDARY OUTCOMES:
Mortality at 28 days | 28 days
  To determine the 28 day mortality from patients with severe AH and spontaneous liver function improvement treated with Methylprednisolone or placebo
Incidence of infections during the study period (90 days) | 90 days
  To determine the incidence of infections during the 90 day study period in corticosteroid-treated compared to placebo-treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Moreno, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- CUB Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucey MR, Mathurin P, Morgan TR. Alcoholic hepatitis. N Engl J Med. 2009 Jun 25;360(26):2758-69. doi: 10.1056/NEJMra0805786. No abstract available. PMID 19553649
- [Background] Maddrey WC, Boitnott JK, Bedine MS, Weber FL Jr, Mezey E, White RI Jr. Corticosteroid therapy of alcoholic hepatitis. Gastroenterology. 1978 Aug;75(2):193-9. PMID 352788
- [Background] Mathurin P, Mendenhall CL, Carithers RL Jr, Ramond MJ, Maddrey WC, Garstide P, Rueff B, Naveau S, Chaput JC, Poynard T. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis (AH): individual data analysis of the last three randomized placebo controlled double blind trials of corticosteroids in severe AH. J Hepatol. 2002 Apr;36(4):480-7. doi: 10.1016/s0168-8278(01)00289-6. PMID 11943418
- [Background] Carithers RL Jr, Herlong HF, Diehl AM, Shaw EW, Combes B, Fallon HJ, Maddrey WC. Methylprednisolone therapy in patients with severe alcoholic hepatitis. A randomized multicenter trial. Ann Intern Med. 1989 May 1;110(9):685-90. doi: 10.7326/0003-4819-110-9-685. PMID 2648927
- [Background] European Association for the Study of Liver. EASL clinical practical guidelines: management of alcoholic liver disease. J Hepatol. 2012 Aug;57(2):399-420. doi: 10.1016/j.jhep.2012.04.004. Epub 2012 May 26. No abstract available. PMID 22633836
- [Background] O'Shea RS, Dasarathy S, McCullough AJ; Practice Guideline Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Alcoholic liver disease. Hepatology. 2010 Jan;51(1):307-28. doi: 10.1002/hep.23258. No abstract available. PMID 20034030
- [Background] Mathurin P, O'Grady J, Carithers RL, Phillips M, Louvet A, Mendenhall CL, Ramond MJ, Naveau S, Maddrey WC, Morgan TR. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis: meta-analysis of individual patient data. Gut. 2011 Feb;60(2):255-60. doi: 10.1136/gut.2010.224097. Epub 2010 Oct 12. PMID 20940288
- [Background] Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, Downs N, Gleeson D, MacGilchrist A, Grant A, Hood S, Masson S, McCune A, Mellor J, O'Grady J, Patch D, Ratcliffe I, Roderick P, Stanton L, Vergis N, Wright M, Ryder S, Forrest EH; STOPAH Trial. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med. 2015 Apr 23;372(17):1619-28. doi: 10.1056/NEJMoa1412278. PMID 25901427